CLINICAL TRIAL: NCT04673890
Title: Improving Cancer Survival and Reducing Treatment Variations With Protocols for Emergency Care (ICARE)
Brief Title: Improving Cancer Survival and Reducing Treatment Variations With Protocols for Emergency Care
Acronym: ICARE
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Heather Prendergast, Professor, University of Illinois at Chicago
Other Study IDs: 2020-0170; 6U48DP006392 (NIH)
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Significant challenges and gaps remain in navigating transitions between acute care and outpatient care for many cancer survivors. This study underscores 1) implementation of Emergency Department (ED) risk-stratified treatments protocols that standardize patient care and would allow for rapid re-assessment and access to specialist care with well-coordinated cancer care plans, and 2) the significant numbers of minority cancer survivors seeking episodic care in the ED that are at increased risk of not receiving recommended post cancer treatment surveillance.

DETAILED DESCRIPTION:
The over-arching goal of this study is to develop a portable model for ED cancer treatment guidelines and management using evidence based protocols in a population at high risk for poor cancer -related outcomes by identifying & overcoming specific barriers to enhanced survivorship. Based on the demographics of ED population (currently, 70% racial/ethnic minorities), the majority of participants will be underrepresented (African-American and Hispanic) and low-income individuals. The investigators propose a feasibility study of 150 patients in the ED over a 1 year period.

The specific aims are:

Aim 1: Evaluate the effectiveness of ED Risk-Stratified, Evidence-Based Treatment protocols on the primary outcome of ED utilization rates and subsequent acute inpatient admissions at 6 -months post-intervention.

Aim 2: Evaluate the effectiveness of an ED-based Cancer Patient Navigator on the secondary outcomes of patient engagement and primary care engagement at 6 -months post-intervention.

Aim 3: Examine barriers and facilitators to compliance for cancer survivorship recommendations that occur in an ED setting at 6-months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor (has had cancer in their lifetime, and is currently disease-free)
* Verbal fluency in English or Spanish
* Age 18-75 years

Exclusion Criteria:

* Unable to verbalize comprehension of study or impaired decision making (e.g., dementia)
* Plans to move from Chicago area within the next year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient recruitment will be completed in the UI Health ED with ED patients who have had a cancer in their lifetime.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
ED utilization rate | 6 months from study entry
  Emergency department utilization over 6 month period
Mortality | 30 days from study entry
  Mortality due to deep vein thrombosis/pulmonary embolism, due to sepsis, and overall mortality
Mortality | 90 days from study entry
  Mortality due to deep vein thrombosis/pulmonary embolism, due to sepsis, and overall mortality
Mortality | 1 year from study entry
  Mortality due to deep vein thrombosis/pulmonary embolism, due to sepsis, and overall mortality

SECONDARY OUTCOMES:
Admission and Readmission rate | 6 months from study entry
  all cause, and related to sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prendergast, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh GK, Jemal A. Socioeconomic and Racial/Ethnic Disparities in Cancer Mortality, Incidence, and Survival in the United States, 1950-2014: Over Six Decades of Changing Patterns and Widening Inequalities. J Environ Public Health. 2017;2017:2819372. doi: 10.1155/2017/2819372. Epub 2017 Mar 20. PMID 28408935
- [Background] Moore JX, Akinyemiju T, Bartolucci A, Wang HE, Waterbor J, Griffin R. A prospective study of cancer survivors and risk of sepsis within the REGARDS cohort. Cancer Epidemiol. 2018 Aug;55:30-38. doi: 10.1016/j.canep.2018.05.001. Epub 2018 May 25. PMID 29763753
- [Background] Connolly GC, Francis CW. Cancer-associated thrombosis. Hematology Am Soc Hematol Educ Program. 2013;2013:684-91. doi: 10.1182/asheducation-2013.1.684. PMID 24319253
- [Background] Naess IA, Christiansen SC, Romundstad P, Cannegieter SC, Rosendaal FR, Hammerstrom J. Incidence and mortality of venous thrombosis: a population-based study. J Thromb Haemost. 2007 Apr;5(4):692-9. doi: 10.1111/j.1538-7836.2007.02450.x. PMID 17367492
- [Derived] Prendergast HM, Khosla S. Lessons learned about policymaking: Moving an emergency department-initiated screening protocol to systemwide input in the development and implementation process. Acad Emerg Med. 2023 Jun;30(6):683-686. doi: 10.1111/acem.14672. Epub 2023 Feb 24. No abstract available. PMID 36707976